CLINICAL TRIAL: NCT05943093
Title: Expression of Long Non-Coding RNA H19 in Acute Lymphoblastic Leukemia
Brief Title: H19 in Acute Lymphoblastic Leukemia.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Refaat Ibrahim Ismail, resident doctor, Assiut University
Other Study IDs: PCR in acute leukemia
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Acute Lymphoid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALL patients
- control group free from the disease

SUMMARY:
* Study the expression level of H19 gene in the samples from ALL patients by real-time PCR.
* Correlate the expression level of H19 gene with the clinical presentation and laboratory data of those patients.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is the most common cancer affecting children and adolescents (Zeng XL et al, 2023). ALL is a haematological malignancy characterized by the malignant clonal expansion of lymphoid hematopoietic precursors (Hong Z et al, 2021). It arises from B- or T-lineage lymphoid progenitors: B-cell-precursor ALL (B-ALL) and T-cell ALL (T-ALL) (Brady SW et al., 2022). Rrelapse in ALL is the fundamental cause of treatment failure in 15-20% of patients (Hulleman E et al, 2009). Therefore, the exploration of novel functional molecules that play a role in ALL pathogenesis could be effective therapeutic targets for this disease (Asadi M et al, 2023).

Long non-coding RNAs (lncRNAs) are non-protein coding transcripts longer than 200 nucleotides (Kopp F et al, 2018). H19 was the first lncRNA to be discovered and submitted for genomic imprinting (Yoshimura H et al, 2018). It has a role in embryogenesis and tumorigenesis (Yoshimura H et al, 2014). It also has an indispensable role in enhancing cell proliferation, differentiation, migration, invasion, and chemo resistance (Li Y et al, 2020). Recent evidence has shown that H19 is an oncogene and is overexpressed in breast, liver, endometrial, lung, cervical, and esophageal cancers (Asadi M et al, 2023). A similar pattern of H19 expression was observed in various types of leukemias, including chronic myeloid leukemia (CML) (Morlando M et al, 2015) and acute myeloid leukemia (AML) (Zhang Tj et al, 2018).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ALL patients.

Exclusion Criteria:

- 1-Presence of other haematological disorders, history of other malignancies or relapsed ALL.

2-Patients under chemotherapy or radiotherapy.

Ages: 2 Months to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: newly diagnosed ALL patients
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
- Study the expression level of H19 gene in the samples from ALL patients by real-time PCR. | baseline

SECONDARY OUTCOMES:
Correlate the expression level of H19 gene with the clinical presentation and laboratory data of those patients. | baseline

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36680478/